CLINICAL TRIAL: NCT01794936
Title: VTI Doppler Probe For Robotic Surgery
Brief Title: Pilot Study of VTI Doppler Probe Use to Identify Neurovascular Bundle During Prostate Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the institution
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: AAAF3321
Record Dates: First submitted 2013-02-09; First posted 2013-02-20 (Estimated); Results first posted 2016-04-22 (Estimated); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer; Nerve Sparing Prostatectomy
Keywords: Prostate cancer; Nerve Sparing Prostatectomy; VTI Probe
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VTI Probe (Experimental): During robotic-assisted laparoscopic prostatectomy, the VTI Doppler probe (test) will utilized to measure blood blow within the neurovascular bundles. This is to be completed after the bladder neck and seminal vesicles are identified and dissected. To use the probe, the assistant surgeon will place the Doppler probe within the abdomen and systematically move it cephalad along the lateral prostate pedicles to identify NVB vessels. The Doppler flow in these regions will be quantified as arterial (strong) flow, venous (minimal) flow or no flow. The procedures will proceed by dissecting the lateral margin of prostate step by step up to the gland's apex. Blood loss and the time required to identify and dissect the NVB will be recorded.
  Interventions: Device: VTI Probe
- Non-Probe (No Intervention): Patients randomized to not receive probe evaluation.

INTERVENTIONS:
Device: VTI Probe — The VTI 20 MHz microvascular Laparoscopic Doppler System is a blood flow detector that compensates for the loss of tactile sensation during laparoscopic procedures by eliminating misunderstandings related to surrounding vascular anatomy. The system's sterile doppler probes fit through standard 5mm ports, making it easy to use with no special training required.
  Arms: VTI Probe

SUMMARY:
This study is designed to evaluate the use of a disposable laparoscopic Doppler probe in robotic assisted prostatectomies. The Vascular Technology, Inc. (VTI) laparoscopic probe is simply a sterile, disposable Doppler probe that can be inserted through a laparoscopic trocar and placed on structures to determine if there is vascular flow demonstrating an audible pulse. During robotic-assisted prostatectomy, identification of vasculature is critical in order to prevent hemorrhage and effectively treat the underlying pathology. The investigators routinely utilize a combined Doppler ultrasound laparoscopic probe to identify vasculature during renal surgery, but Doppler ultrasound usage has not been adopted for prostatic surgery.

From a mechanical standpoint, these combination probes differ from the VTI probe in that they are approximately 2 times the diameter of the VTI probe, and the portion of the probe utilized for imaging much longer and on the side of the device. The VTI probe is much narrower, and the portion of the probe utilized for vessel identification is at the tip of the probe. For robotic-assisted prostatectomy, patients will be randomized to VTI laparoscopic Doppler System to identify pedicles and neurovascular bundles (NVB) or to robotic-assisted laparoscopic prostatectomy with no Doppler probe, which is the current standard of care.

DETAILED DESCRIPTION:
The VTI Laparoscopic Doppler System is a blood flow detector that compensates for the loss of tactile sensation during laparoscopic procedures by helping the surgeon to identify vascular anatomy before it is visible to the eye. The system's sterile doppler probes fit through standard 5mm ports. It is simple to use and no special training is required. This study is designed to evaluate the use of the VTI (Nashua, NH) 20 megahertz (MHz) Microvascular Doppler probe in laparoscopic urological surgery.

Patients will take a preoperative sexual health inventory for men (SHIM) questionnaire. The investigators will then assess presence or absence of arterial and venous blood flow, in real-time during surgery. Additionally, the investigators will evaluate the safety of Doppler probe use, the surgical margin status on final pathology, and the post-operative erectile function of the patients with a followup SHIM questionnaire (to be performed 3 months after surgery). Finally, the robotic surgeon will document whether or not our original surgical plan was changed or remained the same after the Doppler use.

ELIGIBILITY:
Inclusion Criteria:

* All patients must be 18 years of age or older and be able to read, understand and sign consent.
* Any patient undergoing robotic assisted laparoscopic prostatectomy (RALP)
* Any patient without moderate or severe erectile dysfunction (SHIM less than 15) undergoing bilateral or unilateral nerve-sparing RALP is eligible for this procedure.

Exclusion Criteria:

* Patients undergoing a non nerve-sparing RALP will be excluded from this study
* Those who receive a baseline SHIM score less than 15

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ketan Badani, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The principal investigator has left the institution. Attempts to contact the PI have been unsuccessful. Columbia will never have access to the data. Thus, data will not be analyzed. The only information available is the number of participants who started and completed the study, which was last reported to and approved by the IRB in February 2012.
Groups:
- VTI Probe or Non-Probe: Data per arm is not available. Columbia will never have access to this data.
Period: Overall Study
Arm/Group | VTI Probe or Non-Probe
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | VTI Probe or Non-Probe
Number analyzed (Participants) | 9
Age, Customized [Number; unit: participants]
  18 years and older | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in SHIM Score (Score of Erectile Function) Following Surgery
Description: Patients are to be evaluated for erectile function at 8 month post-operative visit using validated SHIM questionnaire.
Time Frame: 8 months post-operative follow-up
Population: The principal investigator has left the institution. Attempts to contact the PI have been unsuccessful. Columbia will never have access to the data. Thus, data will not be analyzed. The only information available is the number of participants who started and completed the study, which was last reported to and approved by the IRB in February 2012.
Arm/Group | VTI Probe or Non-Probe
Number analyzed (Participants) | 0

2. Primary Outcome: Prevalence of Intra-operative Complications
Description: Investigators will evaluate whether any intra-operative complications resulted from the use of the VTI probe to assess safety. Specifically, this time frame is limited from the induction of anesthesia through the completion of the surgical procedure (typically ~2-3 hours)
Time Frame: During surgical procedure itself (~2-3 hours)
Population: as for outcome 1
Arm/Group | VTI Probe or Non-Probe
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The principal investigator has left the institution. Attempts to contact the PI have been unsuccessful. Columbia will never have access to the data. Thus, data will not be analyzed. The only information available is the number of participants who started and completed the study, which was last reported to and approved by the IRB in February 2012.
Arm/Group | VTI Probe or Non-Probe
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No